CLINICAL TRIAL: NCT02930096
Title: Study of the Effect of the Supine Position at Brain Velocities in Noncerebro - Injured Patient
Acronym: D-Velocity
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D-Velocity
Record Dates: First submitted 2016-10-04; First posted 2016-10-12 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pulsatility index mesured with doppler ultrasound

SUMMARY:
To evaluate the pulsatility index changes after setting supine position in non brain- injured patient under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old, maximum 45 years old for men and 55 years old for women.
* surgery with supine position.

Exclusion Criteria:

* refusal to participate
* failure of measurement brain velocity
* Penthotal or de kétamine before measurment
* Cardiac or pulmonary desease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient who need a surgery in supine position and who don't have brain injured or pulmonary desease.
  Forty patients over 24 month period were included in the study, after informed consent.
  Pulsatility index is mesured with doppler ultrasound:
  1. before general anesthesia
  2. after general anesthesia in dorsal position
  3. in supine position
  4. in supine position with 15° proclive Evaluation to the pulsatility index changes in theese position
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03

PRIMARY OUTCOMES:
Evaluation the pulsatility index after setting prone position in non brain-injured patient | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- DAHYOT FIZELIER Claire, Poitiers, France